CLINICAL TRIAL: NCT05453669
Title: Clinical Study of the Efficacy of CD19-CAR-DNT Cells in the Treatment of Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Clinical Study of the Efficacy of CD19-CAR-DNT Cells in the Treatment of Relapsed/Refractory B-cell NHL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Ruijiamei Biotechnologies, Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2022000371
Record Dates: First submitted 2022-06-28; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
Keywords: r/r B-NHL ,Cell therapy
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-CAR-DNT cells (Experimental): 9 patientsare planned to be enrolled in the dose-escalation trial (1×10^6 CD19-CAR-DNT cells/kg, 3×10^6 CD19-CAR-DNT cells/kg, 9×10^6 CD19-CAR-DNT cells/kg) and 3 patients in the dose-expansion trial.
  Interventions: Biological: CD19-CAR-DNT cells

INTERVENTIONS:
Biological: CD19-CAR-DNT cells — Lentiviral vector-transducted DNT cells to express anti-CD19 CAR. Prior to cellular infusion, each patient received cyclophosphamide and fludarabine lymphodepleting chemotherapy.

SUMMARY:
To evaluate the safety and tolerability of CD19-CAR-DNT cells infusion in subjects with relapsed/refractory B-cell non-Hodgkin's Lymphoma

DETAILED DESCRIPTION:
This is an open, single-arm, single-dose, dose-escalation and dose-expansion clinical trial designed to evaluate the maximum tolerated dose of CD19-CAR-DNT cells, the safety, the preliminary efficacy and the pharmacokinetic profile of CD19-CAR-DNT cells in vivo after infusion in clinical studies. 9 patients are planned to be enrolled in the dose-escalation trial (1×10^6 CD19-CAR-DNT cells/kg, 3×10^6 CD19-CAR-DNT cells/kg, 9×10^6 CD19-CAR-DNT cells/kg) and 3 patients in the dose-expansion trial. The primary endpoints are DLT, MTD, and the incidence of abnormalities in AE/SAE/AESI/laboratory tests/electrocardiograms/vital signs.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an ICF and expect to complete the study procedures for follow-up examinations and treatment.
2. Aged 18 to 75 years (including cut-offs), regardless of gender
3. A diagnosis of B-cell non-Hodgkin's lymphoma confirmed by cytology or pathological histology according to WHO 2016 criteria, including pathologically confirmed diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), transformed follicular lymphoma (TFL) and high-grade B-cell lymphoma (HGBCL).
4. Relapsed/refractory B-cell non-Hodgkin's lymphoma, provided one of the following conditions is met:

   * Subjects with B-cell non-Hodgkin's lymphoma who have failed at least second-line regimens (including relapse, non-remission, progression) and have received a standardised regimen of anti-CD20 monoclonal antibodies (except CD20-negative) and anthracyclines;
   * Relapse after autologous haematopoietic stem cell transplantation;
   * Primary resistance: induction with 2 courses of anti-CD20 monoclonal antibody-based immunochemotherapy at the time of first treatment, the best curative effect assessed as stable disease or disease progression.
5. ECOG score 0 to 1.
6. The presence of a measurable lesion that meets one of the following criteria:

   * The long axis of the lymph node lesion exceeds 15 mm in length (the short axis is measurable);
   * The long and short axes of the extralymph node lesion exceed 10 mm in length.
7. Appropriate organ function, with laboratory results within 7 days prior to lymphatic clearance chemotherapy meeting the following criteria.

   * Glutathione aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN)
   * Glutamic aminotransferase (ALT) ≤ 3 times ULN.
   * Total bilirubin ≤ 1.5 times ULN, unless the subject has documented Gilbert syndrome. Subjects with Gilbert-Meulengracht syndrome with total bilirubin ≤ 3.0 times ULN and direct bilirubin ≤ 1.5 times ULN may be included.
   * Serum creatinine ≤ 1.5 times ULN or a creatinine clearance ≥ 60 ml/min.
   * Haemoglobin ≥ 60 g/L or haemoglobin maintained at that level following transfusion.
   * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L.
   * A platelet count ≥ 30 x 10^9/L or a platelet count maintained at that level following a platelet transfusion
   * Left ventricular ejection fraction (LVEF) ≥ 45%.
8. Female subjects with of childbearing potential should have a negative pregnancy test during the screening period. Any male and female subjects of childbearing potential must agree to use an effective contraception method for at least six months from the time that they sign the informed consent form until the end of the cell infusion. Female subjects without childbearing potential (meeting at least 1 of the following criteria) is described below.

   * Have undergone a hysterectomy or bilateral oophorectomy
   * Medically recognised ovarian failure.
   * Medically recognised as post-menopausal (at least 12 consecutive months of menopause without pathological or physiological cause).

Exclusion Criteria:

1. Other malignancies within 5 years prior to screening, except adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer, post-radical localized prostate cancer, post-radical ductal carcinoma in situ, and post-radical thyroid cancer
2. Any unstable systemic disease: including but not limited to active infection (other than local infection), unstable angina, cerebrovascular accident or transient ischaemia (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), New York Heart Association class III or IV cardiac insufficiency, refractory hypertension (refractory hypertension is defined as blood pressure that has not reached standard after >1 month of reasonably tolerable treatment with ≥3 antihypertensive drugs (including diuretics) at adequate doses based on lifestyle improvement or blood pressure that is not effectively controlled with ≥4 antihypertensive drugs), severe cardiac arrhythmias requiring pharmacologic treatment, hepatic arrhythmias, liver diseases, kidney diseases or metabolic disorders.
3. Patients with B-cell non-Hodgkin's lymphoma with active central nervous system invasion.
4. Patients with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titres not within the normal reference range, positive hepatitis C virus (HCV) antibody and peripheral blood HCV RNA ,positive for human immunodeficiency virus (HIV), or positive for cytomegalovirus (CMV) DNA, or positive syphilis test.
5. Active or uncontrolled infections requiring systemic treatment (except simple urinary tract infections or upper respiratory tract infections).
6. Subjects who are receiving systemic steroids prior to screening and who are judged by the investigator to require long-term treatment with systemic steroids during the treatment period (except for inhaled or topical use).
7. Previous organ transplantation or preparation for organ transplantation (except for haematopoietic stem cell transplantation)
8. Persons with acute/chronic Graft-vs-Host Disease (GvHD)
9. Patients have received a haematopoietic stem cell transplant within 2 months prior to screening
10. Patients have received CAR-T therapy or other gene-modified cell therapy prior to enrolment
11. Active neurological autoimmune or inflammatory diseases (e.g. Guillain-Barre Syndrome (GBS), Amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular disease (e.g. cerebral oedema, Posterior Reversible Encephalopathy Syndrome (PRES)). Encephalopathy Syndrome (PRES)).
12. Patients with a life expectancy of less than 3 months
13. Patients have been involved in other clinical studies within 3 months prior to screening.
14. Patients, in the judgement of the investigator and/or clinical criteria, are contraindicated to any study procedure or have other medical conditions that may place them at unacceptable risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of CD19-CAR-DNT Cell Therapy for Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
MTD | Up to 28 days
  MTD was the highest dose for DLT in ≤1/6 subjects
Incidence of abnormalities | Up to 28 days
  Incidence of abnormalities in AE/SAE/AESI/laboratory tests/electrocardiograms/vital signs.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) indicator (Cmax) | Up to 90 days
  The peak concentration of CD19-CAR-DNT cells amplified in the peripheral blood (Cmax, detected by qPCR).
Pharmacokinetics (PK) indicator (AUC) | Up to 90 days
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the area under the curve (AUC). (AUC, detected by qPCR).
Pharmacokinetics (PK) indicator (Tmax) | Up to 90 days
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the peak plasma time (Tmax). Tmax is defined as the time to reach the highest concentration (Tmax, detected by qPCR).
Pharmacokinetics (PK) indicator (T1/2) | Up to 90 days
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the elimination half-life in hours (T1/2). T1/2 is defined as the time point when the concentration of CD19-CAR-DNT reaches half of maximum in a patient's peripheral blood (T1/2, detected by qPCR).
Overall Response Rate | Up to 2 years
  The proportion of CR or PR patients as assessed by investigators based on Lugano 2014 Response Assessment
Disease Control Rate | Up to 2 years
  The percentage of PR, CR and SD patients in the total patient population
Duration of Response | Up to 2 years
  The time from the start of the first assessment of CR or PR to the first assessment as disease recurrence or progression or death
Progression Free Survival | Up to 2 years
  The length of time that a participant's disease did not progress during or after CD19-CAR-DNT treatment.
Overall Survival | Up to 15 years
  From the date of entry into the clinical study until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, MD, PhD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao X, Liu H, Qiu X, Chen P, Li X, Wang D, Song G, Cheng Y, Yang L, Qian W. CD19-CAR-DNT cells (RJMty19) in patients with relapsed or refractory large B-cell lymphoma: a phase 1, first-in-human study. EClinicalMedicine. 2024 Feb 29;70:102516. doi: 10.1016/j.eclinm.2024.102516. eCollection 2024 Apr. PMID 38444429